CLINICAL TRIAL: NCT06734585
Title: A Comparison Between Gilteritinib in Phase 3 Trials Versus Real-World External Comparator Cohort of Relapsed/Refractory (R/R) FLT3m+ Acute Myeloid Leukemia (AML) Patients After Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Using Gilteritinib to Keep People With Acute Myeloid Leukemia Cancer-free After a Stem Cell Transplant
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Singapore Pte. Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 2215-MA-3574
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: Gilteritinib; Xospata; Relapsed or refractory FLT3m+ Acute Myeloid Leukemia (AML); Hematopoietic Stem Cell Transplantation (HSCT); Best Supportive Care
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — gilteritinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- External Comparator: Participants with R/R Feline McDonough Sarcoma-like Tyrosine Kinase 3 Mutation (FLT3)+AML who underwent HSCT after achieving any type of complete remission (CR) and who received best supportive care after HSCT.
- Gilteritinib: Participants with R/R FLT3+AML who were enrolled in the ADMIRAL and COMMORDORE phase 3 studies that resumed gilteritinib after HSCT to maintain remission.
  Interventions: Drug: Gilteritinib

INTERVENTIONS:
Drug: Gilteritinib — tablet, oral
  Other Names: ASP2215; XOSPATA®
  Groups: Gilteritinib

SUMMARY:
People with acute myeloid leukemia (AML) are usually treated with chemotherapy. When the cancer comes back (relapse) the next treatment is usually a stem cell transplant. Some people with AML have a changed FLT3 gene which causes leukemia cells to grow faster. This means their cancer may come back more quickly after treatment.

Gilteritinib is approved in many countries to treat people with AML with the changed FLT3 gene whose cancer has come back or have not responded to previous treatment. In some countries, more studies are needed to approve gilteritinib for use.

This study is about people with AML with the changed FLT3 gene. The main aim was to learn if gilteritinib improves how long people stay cancer-free (in remission) after a stem cell transplant. To do this, 2 groups were compared. 1 group were given gilteritinib after a stem cell transplant. This happened in previous studies called the ADMIRAL study and COMMODORE study. The other group received standard of care after their stem cell transplant. They did not receive gilteritinib after their stem cell transplant.

In this study, information about the people who received standard of care after their stem cell transplant will be collected. This study is about collecting information only. The study sponsor (Astellas) will not provide any treatment.

Information will be collected from the people's medical records between 01 Jan 2015 and 31 Dec 2022. The study doctors will collect information from the first relapse, during and after the stem cell transplant. Then, they will record when any of the following happened after the stem cell transplant: the person passed away, their cancer came back, they decided to leave the study or could not be contacted.

ELIGIBILITY:
Inclusion Criteria:

Gilteritinib Group

* Patients from ADMIRAL and COMMODORE phase 3 studies that resumed gilteritinib after HSCT to maintain remission

External Comparator Group

* Patient with a diagnosis of AML according to World Health Organization (WHO) classification
* Patient with positive either FLT3-Internal Tandem Duplications (ITD) or FLT3- Tyrosine Kinase Domain (TKD) genetic testing or re-testing
* Patient with pre-defined first R/R AML at enrollment:

  * Refractory to first-line AML therapy is defined as patient not achieving CR/Complete Remission with Incomplete Hematologic Recovery (CRi)/Complete Remission with Incomplete Platelet Recovery (CRp) under initial therapy. A patient eligible for standard therapy must receive at least 1 cycle of an anthracycline containing induction block in standard dose for the selected induction regimen. A patient not eligible for standard therapy must have received at least 1 complete block of induction therapy seen as the optimum choice of therapy to induce remission for this patient.
  * Relapsed after first-line AML therapy. First-line AML therapy is defined as (all criteria must be met): Patient achieved a CR/CRi/CRp (as defined by International Working Group criteria) and Initial AML therapy must have consisted of up to 2 induction blocks with or without consolidation or maintenance, with or without transplantation
* Patient underwent allogenic HSCT upon R/R AML diagnosis
* Patient who was alive at 90 days post-HSCT and:

  * Patient had successful engraftment as demonstrated by absolute neutrophil count (ANC) ≥ 500/mm3 and platelets ≥ 20000/mm3 without transfusions
  * Patient did not have grade 3 or above acute GvHD
  * Patient was in any type of CR
* Patient who received best supportive care after HSCT; Best supportive care refers to treatment(s) patients received in CR after HSCT and remained in CR when given the intervention. This may include prophylactic intrathecal chemotherapy, cranial radiation, and donor lymphocyte infusion as part of the HSCT treatment plan.

Exclusion Criteria:

External Comparator Group

* Eastern Cooperative Oncology Group (ECOG) ≥ 2
* Patients who received midostaurin, sorafenib, gilteritinib, or venetoclax, or chemotherapy post-HSCT as maintenance therapy prior to index date
* Patient diagnosed with acute promyelocytic leukemia
* Enrollment in drug interventional post-HSCT AML clinical trials during study period
* Critical information is not available for abstraction; Critical information includes FLT3m+confirmation, R/R confirmation, transplantation outcomes (e.g., any type of CR, any grade 3 or above GvHD) at 90 days post-HSCT

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The external comparator group will include participants with R/R FLT3+AML who underwent HSCT after achieving any type of CR and who received best supportive care after HSCT. Data for the gilteritinib group will be obtained from a subgroup of ADMIRAL and COMMODORE phase 3 studies that resumed gilteritinib after HSCT to maintain remission.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2025-01-09 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Relapse Free Survival (RFS) | 12 months after index date (90 days post-HSCT)
  RFS is defined as the time from index date to the date of relapse or the date of death from any cause, whichever comes first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 24 months after index date (90 days post-HSCT)
  OS is defined as time from the index date until the date of death from any cause.
Graft-versus-host disease (GvHD)-free relapse-free survival (GFS) | 12 months after index date (90 days post-HSCT)
  GFS is defined as the time from the index date to the date of grades III to IV acute GvHD, chronic GvHD requiring systemic treatment, cytogenetic or hematologic relapse, and death from any cause after HSCT.
Cumulative Incidence of Relapse | Up to 24 months
  Cumulative incidence of relapse is defined as the time from the index date to the date of first relapse, with non-relapse related death (or death in complete remission) being the competing risk.

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Singapore Pte. Ltd.
Locations (18):
- Australia (2):
  - AU61001, Melbourne
  - AU61002, Melbourne
- Brazil (4):
  - BR55004, Fortaleza
  - BR55002, Porto Alegre
  - BR55001, São Paulo
  - BR55003, São Paulo
- China (3):
  - CN86003, Shanghai
  - CN86004, Suzhou
  - CN86001, Tianjin
- HK852001, Hong Kong, Hong Kong
- South Korea (5):
  - KR82004, Busan
  - KR82005, Gwangju
  - KR82001, Seoul
  - KR82002, Seoul
  - KR82003, Seoul
- Taiwan (3):
  - TW88603, Taichung
  - TW88602, Tainan
  - TW88601, Taipei

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.